CLINICAL TRIAL: NCT01152775
Title: Evaluation of the Use of Multimedia to Enhance Patient and Family Understanding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. David Fleiszer, 2) Associate Professor of Surgery, McGill University, Faculty of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-269-PSY
Record Dates: First submitted 2010-06-17; First posted 2010-06-29 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: The Role of Multimedia on Retention and Comprehension of Key Concepts for Surgical Options in Newly Diagnosed Breast Cancer Patients.
Keywords: partnered surgical decision-making; impact of multimedia-based teaching; patient education; understanding and retention by patients

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Media (Placebo Comparator): Sixty participants will be randomized into one of two cohorts: 1. No media 2. Yes media
  Interventions: Other: No Media
- Yes Media Newly Diagnosed Breast Cancer Pts (Experimental): Sixty participants will be randomized into one of two cohorts: 1. No media 2. Yes media
  Interventions: Other: This group of patients will be exposed to multimedia

INTERVENTIONS:
Other: This group of patients will be exposed to multimedia — This group of patients will be exposed to multimedia
  Arms: Yes Media Newly Diagnosed Breast Cancer Pts
Other: No Media — This group will not be exposed to multimedia
  Arms: No Media

SUMMARY:
This study will investigate the potential impact of arts-informed, technology-based patient education material, and specifically, the role of multimedia imagery on patient comprehension, perceived satisfaction, anxiety levels, and informed decision-making.

DETAILED DESCRIPTION:
Based on an inter-professional approach to support a new role in patient care, this research addresses both literacy and health literacy issues within the context of current challenges to healthcare delivery and associated fragmentation in continuity of care. Patient education is a key component in the delivery of comprehensive care and it is the potential for on-line patient education that provides the basis for research.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be used: Participants must be:

1. Newly diagnosed breast cancer patients
2. A minimum age of 18 years or older
3. Able to read and write in English and/or French
4. Have a confirmed diagnosis of any of the following:

   1. Infiltrating ductal carcinoma
   2. Ductal carcinoma in situ (Grade III)
   3. Lobular carcinoma in situ (Grade III)
   4. Infiltrating lobular carcinoma
5. Have access to, and the ability to use, a computer

Exclusion Criteria:

* The following criteria will be reasons for exclusion from the study:

  1. The participant has a serious psychiatric or cognitive impairment that would prevent the patient from completing the study requirements.
  2. The participant has a previous history of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Concept Grid | 1 year
  A likert scale measuring the comprehension and retention of key concepts in the research study.

SECONDARY OUTCOMES:
DCS Conflict Scale | 1 year
  Traditional Decision Conflict Scale - The decisional conflict scale measures personal perceptions of: a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction.
Anxiety Scale - A.S. Zigmond and R.P. Snaith | 1 year
  A self-assessment scale that has been developed and found to be a reliable instrument for detecting states of depression and anxiety in the setting of a hospital medical outpatient clinic. This questionnaire is designed to help the doctor know how you feel.
The Hospital Anxiety and Depression (HAD) Scale | 1 year
  The Hospital Anxiety and Depression (HAD) rating scale is a commonly used questionnaire. It is a screening questionnaire for psychiatric disorders.
Interactive Patient Education Oncology Module | 1 year
  We would like to know if the module helped the patient understand their disease and their available treatment options. It is a questionnaire to obtain feedback on its overall design.

CONTACTS AND LOCATIONS:
Overall Officials: David Fleiszer, M.D.C.M., F.R.C.S (C)., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Nancy Posel, N. DIA, M.Ed, PhD, Study Director — McGill University; Dianne Bateman, PhD, Study Chair — McGill University
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Cedars Breast Clinic, Montreal, Quebec
  - Myrna Cabaluna, Manager, MUHC Education Portfolio, Montreal, Quebec

REFERENCES:
- [Background] del Carmen MG, Joffe S. Informed consent for medical treatment and research: a review. Oncologist. 2005 Sep;10(8):636-41. doi: 10.1634/theoncologist.10-8-636. PMID 16177288
- [Background] Etchells E, Sharpe G, Walsh P, Williams JR, Singer PA. Bioethics for clinicians: 1. Consent. CMAJ. 1996 Jul 15;155(2):177-80. PMID 8800075
- [Result] Beamond BM, Beischer AD, Brodsky JW, Leslie H. Improvement in surgical consent with a preoperative multimedia patient education tool: a pilot study. Foot Ankle Int. 2009 Jul;30(7):619-26. doi: 10.3113/FAI.2009.0619. PMID 19589307
- [Result] Patel V, Aggarwal R, Kinross J, Taylor D, Davies R, Darzi A. Improving informed consent of surgical patients using a multimedia-based program?: results of a prospective randomized multicenter study of patients before cholecystectomy. Ann Surg. 2009 Mar;249(3):546-7; author reply 547-8. doi: 10.1097/SLA.0b013e31819abeb1. No abstract available. PMID 19247056
- [Result] Eggers C, Obliers R, Koerfer A, Thomas W, Koehle K, Hoelscher AH, Bollschweiler E. A multimedia tool for the informed consent of patients prior to gastric banding. Obesity (Silver Spring). 2007 Nov;15(11):2866-73. doi: 10.1038/oby.2007.340. PMID 18070779
- [Result] Ryhanen AM, Siekkinen M, Rankinen S, Korvenranta H, Leino-Kilpi H. The effects of Internet or interactive computer-based patient education in the field of breast cancer: a systematic literature review. Patient Educ Couns. 2010 Apr;79(1):5-13. doi: 10.1016/j.pec.2009.08.005. Epub 2009 Sep 9. PMID 19744817
- [Result] Sandberg EH, Sharma R, Wiklund R, Sandberg WS. Clinicians consistently exceed a typical person's short-term memory during preoperative teaching. Anesth Analg. 2008 Sep;107(3):972-8. doi: 10.1213/ane.0b013e31817eea85. PMID 18713916